CLINICAL TRIAL: NCT05543135
Title: Aetiology of Asymmetrical Hearing Loss: A Retro-spective Study Thesis Submitted for Partial Fulfillment of Master Degree in Audio-Vestibular Medicine
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Inas Mahmoud Mahrous, resident doctor at audiovestibular unit Qena general hospital, Sohag University
Other Study IDs: Soh-Med-22-07-09
Record Dates: First submitted 2022-09-14; First posted 2022-09-16 (Actual); Last update posted 2022-09-16 (Actual); Status verified 2022-09

CONDITIONS: Asymmetrical Hearing Loss

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- cases: patients with asymmetrical hearing loss
  Interventions: Diagnostic Test: basic audiological evaluation

INTERVENTIONS:
Diagnostic Test: basic audiological evaluation — pure tone audiometry&immitancemetry
  Other Names: CT&MRI

SUMMARY:
Hearing loss maybe: -Symmetrical: in which the severity and pattern of hearing loss are the same in each ear. Or -Asymmetrical: is defined as binaural difference in bone conduction thresholds of >10 dB at two consecutive frequencies or >20 dB at one frequency (0.25-8.0 kHz), Poorer speech perception will often accompany poorer hearing and may be the reason for the patient's presentation .Unilateral or asymmetrical sensorineural hearing loss is important to discern, as it is an important risk factor for auditory nerve tumors (i.e. vestibular schwannoma) which is a life threatening condition, and in such cases further investigation is required (i.e. MRI scan) unless there is a known reason for the asymmetry, Several reports have recommended that further evaluation, especially expensive imaging studies, be conducted to rule out acoustic tumors when AHL is present

ELIGIBILITY:
Inclusion Criteria:

* Age: 6 years old and more.
* Sex: male and female.

Exclusion Criteria:

* Age: less than 6 years old.
* Patients with symmetrical hearing loss.

Min Age: 6 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: all patients with asymmetrical hearing loss with age ranging 6 years old and more.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-09-20 (Estimated); Primary Completion 2023-09 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Asymmetrical hearing loss | 1 year
  asymmetrical hearing loss using basic audiological evalution &imaging

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Dunn CC, Tyler RS, Oakley S, Gantz BJ, Noble W. Comparison of speech recognition and localization performance in bilateral and unilateral cochlear implant users matched on duration of deafness and age at implantation. Ear Hear. 2008 Jun;29(3):352-9. doi: 10.1097/AUD.0b013e318167b870. PMID 18453885
- [Background] Margolis RH, Saly GL. Asymmetric hearing loss: definition, validation, and prevalence. Otol Neurotol. 2008 Jun;29(4):422-31. doi: 10.1097/MAO.0b013e31816c7c09. PMID 18418281
- [Background] Peng AW, Salles FT, Pan B, Ricci AJ. Integrating the biophysical and molecular mechanisms of auditory hair cell mechanotransduction. Nat Commun. 2011 Nov 1;2:523. doi: 10.1038/ncomms1533. PMID 22045002
- [Background] Plack CJ, Barker D, Hall DA. Pitch coding and pitch processing in the human brain. Hear Res. 2014 Jan;307:53-64. doi: 10.1016/j.heares.2013.07.020. Epub 2013 Aug 11. PMID 23938209